CLINICAL TRIAL: NCT04503967
Title: A Phase II Study to Evaluate the Efficacy and Safety of Anlotinib Hydrochloride Combined With Nivolumab in the Treatment of Advanced Gastric Adenocarcinoma and Esophageal Squamous Cell Carcinoma as Second-line or Salvage Chemotherapy
Brief Title: Efficacy and Safety of Anlotinib Hydrochloride Combined With Nivolumab in the Treatment of Gastric and Esophageal Cancer
Acronym: OASIS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Doctor, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OASIS
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Gastric Adenocarcinoma; Esophageal Squamous Cell Carcinoma
Keywords: Gastric Cancer; esophageal cancer; Anlotinib Hydrochloride; Nivolumab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Stomach Neoplasms; Esophageal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Hydrochloride With Nivolumab (Experimental): Anlotinib Hydrochloride Combined With Nivolumab in the second line treatment of Gastric and Esophageal Cancer patients
  Interventions: Drug: Anlotinib Hydrochloride With Nivolumab

INTERVENTIONS:
Drug: Anlotinib Hydrochloride With Nivolumab — Anlotinib Hydrochloride Combined With Nivolumab in the second line Treatment of Gastric and Esophageal Cancer patients

SUMMARY:
Patients with unresectable or metastatic gastric or esophageal cancer, with first-line treatment applied are to be recruited in the study. In the current study, the efficacy and safety of anlotinib hydrochloride combined with nivolumab as second-line or salvage chemotherapy will be evaluated in Chinese patients with advanced gastric adenocarcinoma and esophageal squamous cell carcinoma. 48 patients could provide adequate precision rather than controlling type I&II error.

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteers to participate in the study, signs a consent form, has good compliance, and obeys the follow-up, and is willing and able to follow the protocol during the study.
2. Male or female, aged ≥18 years and ≤75 years.
3. The ECOG PS score is 0 or 1.
4. Histological and/or cytological confirmation of patients with unresectable or metastatic gastric adenocarcinoma or esophageal squamous cell carcinoma.
5. Patients have failed previous first-line standard treatments, have measurable target lesions, and have not received local treatments such as radiotherapy for target lesions (Note: lesions that have previously received radiation therapy cannot be considered target lesions, except that after radiation therapy, clear progress has occurred).
6. At least 4 weeks after previous major surgical and / or radiation therapy (at least 2 weeks after palliative radiotherapy).
7. The use of 0-1 antihypertensive drug can effectively control blood pressure, which is defined as random pre-systolic blood pressure ≤140mmHg, diastolic blood pressure ≤90mmHg, and no antihypertensive drug has been changed within one week before randomization.
8. Appropriate bone marrow reserve, as shown in the blood count of the subject within 7 days before enrollment: hemoglobin ≥90g / L; ANC ≥1.5 × 109 / L; platelet ≥90 × 109 / L (patients have not received blood transfusion or growth factor support within 2 weeks prior blood collection).
9. Appropriate liver function is shown to meet all of the following requirements:

   1. Serum total bilirubin ≤ 1.5 x ULN (Gilbert syndrome patients can be included if the total bilirubin is <3 x ULN, and those with biliary obstruction allow biliary drainage);
   2. serum albumin ≥30g / L;
   3. AST, ALT ≤ 3 x ULN (If liver metastases exist, AST and ALT allow ≤ 5 x ULN).
10. Appropriate renal function demonstrated by all of the following requirements:

    1. Serum creatinine ≤ 1.5 x ULN and creatinine clearance ≥ 50ml/min (using Cockcroft-Gault formula);
    2. Proteinuria <++; if proteinuria is ≥++, 24-hour urine protein must be <2g.
11. INR or prothrombin time (PT) ≤ 1.5 x ULN, APTT ≤ 1.5 x ULN; no history of anticoagulant treatment; investigator judges no high coagulation risk.
12. All acute toxic effects of previous anti-cancer treatment or surgery were all relieved by NCI-CTCAE version 5.0 ≤ 1 (except for hair loss or other toxic effects that the investigator judges to have no risk to the patient's safety).
13. Fertile women must have a negative urine or serum pregnancy test within 7 days before enrollment, and must agree to use effective contraception during the study period and within 6 months after the end of the study period; non-sterile men must agree to use efficient contraception during the study period and within 6 months after the study was completed. Patient agrees to avoid sperm donation during the same time period.
14. Have the ability to act autonomously, have the ability to swallow pills, and have no gastrointestinal diseases that affect oral drug absorption.
15. Agree to provide hematology and histology samples.

Exclusion Criteria:

1. Have undifferentiated or other histological types of gastric or esophageal cancer; evidence of tumor invasion of major blood vessels (including completely adjacent, surrounding, or extending into the main vessel lumen, such as the pulmonary artery or superior vena cava) , and the researcher judges that it is not suitable for enrollment.
2. Patients with active autoimmune disease or a history of autoimmune disease but who may relapse.

   Note: Patients with the following diseases are not excluded and can be entered for further screening:
   1. Controlled Type 1 Diabetes
   2. Hypothyroidism (if only controlled by hormone replacement therapy)
   3. Controlled celiac disease
   4. Skin diseases that do not require systemic treatment (e.g. vitiligo, psoriasis, hair loss)
   5. Any other disease that is not expected to recur without external triggers
3. Any active malignant tumor within 2 years, except for the specific cancer being studied in this trial and cured local recurrent cancer (such as resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ).
4. There is uncontrollable pleural effusion, pericardial effusion, or ascites that need to be drained frequently within 7 days before enrollment (allow effusion cytology to confirm).
5. Patients with gastrointestinal bleeding within two weeks before enrollment, or those at high risk of bleeding as judged by the investigator (Note: fecal occult blood (+) is not an exclusion criterion).
6. Gastrointestinal perforation and / or fistula occurred within 6 months before enrollment.
7. There are many factors that affect oral drug absorption (such as inability to swallow, nausea and vomiting, upper gastrointestinal obstruction, abnormal physiological function, malabsorption syndrome, etc.), which may affect anlotinib hydrochloride absorbers.
8. Weight loss ≥ 20% within 2 months before enrollment.
9. History of the following diseases: interstitial lung disease, non-infectious pneumonia or uncontrollable systemic diseases including diabetes, hypertension, pulmonary fibrosis, acute lung disease, etc.
10. Severe chronic or active infections, including tuberculosis, that require systemic antibacterial, antifungal or antiviral treatment.
11. Known history of HIV infection.
12. Patients with untreated chronic hepatitis B or chronic HBV carriers with hepatitis B virus (HBV) DNA exceeding ULN, or hepatitis C virus (HCV) RNA positive should be excluded. Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable patients with hepatitis B (HBV DNA <ULN), and patients with cured hepatitis C can be selected.
13. Have any of the following cardiovascular risk factors:

    1. Cardiogenic chest pain occurs within ≤ 28 days prior to enrollment, and is defined as moderate pain that limits the daily use of appliance sexual activity.
    2. Symptomatic pulmonary embolism occurred within ≤ 28 days before enrollment.
    3. Acute myocardial infarction occurred within ≤ 6 months before enrollment.
    4. Have any history of heart failure that has reached New York Heart Association Grade III / IV within ≤ 6 months before enrollment, or left ventricular ejection fraction <50%.
    5. Ventricular arrhythmia of grade ≥ 2 occurred within ≤ 6 months before enrollment.
    6. Cerebrovascular accident (CVA) occurred within ≤ 6 months before enrollment
    7. Those with high blood pressure who cannot be controlled well with antihypertensive medications. The symptoms are: systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg (within 3 months).
    8. Significant cardiac conduction abnormalities, including a history of QTc interval prolongation syndrome (QTc interval prolongation> 450 ms) and/or a history of pacemaker implantation.
14. Patients receiving oral or parenteral anticoagulant or thrombolytic treatment for therapeutic purposes during screening and/or during the study should be excluded.
15. The patient has brain metastases or meningeal metastases.
16. People who are allergic to any research medication.
17. Have had an allogeneic stem cell transplant or organ transplant.
18. Corticosteroids (prednisone or similar drugs at doses greater than 10 mg/day are required for ≤ 14 days before enrollment) Equal dose) or other immunosuppressive agents for systemic treatment.

    Note: Patients who are currently or previously using any of the following steroid regimens can be selected:
    1. Adrenaline replacement steroids (prednisone ≤10mg / d or equivalent dose of similar drugs)
    2. Local, ophthalmic, intra-articular, intranasal, and inhaled corticosteroids with minimal systemic absorption.
    3. Short-term (≤ 7 days) use of corticosteroids for prophylaxis (for example, to prevent contrast agent hypersensitivity or antiemetic for specific chemotherapy) or for the treatment of non-autoimmune conditions (such as delayed hypersensitivity caused by contact allergens).
19. Live vaccinations were given within 4 weeks before randomization (Note: seasonal influenza vaccines are usually inactivated vaccines and are allowed. Vaccines used in the nasal cavity are live vaccines and are not allowed).
20. Have received immunotherapy (such as interleukin, interferon, thymosin, etc.) or any experimental treatment within 28 days or 5 half-lives (whichever is shorter, but at least 14 days) before enrollment.
21. Having received anti-PD-1, anti-PD-L1, anti-PD-L2, or any other specific antibody or drug therapy that targets T-cell co-stimulation or checkpoint pathways.
22. For those with a history of uncontrolled epilepsy, central nervous system disease, or mental disorder, it is up to the investigator to determine whether their clinical severity prevents the signing of informed consent or affects the patient's compliance with oral medication.
23. There are potential medical conditions or alcohol/drug abuse or dependence that the investigator believes are not conducive to the administration of the study drug or affect the interpretation of drug toxicity or adverse events.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to 2 years
  The ORR in patients with unresectable or metastatic GC or ESCC patients treated with anlotinib hydrochloride in combination with nivolumab as a second-line or later treatment.

SECONDARY OUTCOMES:
Progression-free survival | up to 2 years
  The PFS was calculated from the initiation of chemotherapy to the date of disease progression or death.
Overall survival | up to 2 years
  Overall survival was measured from the initiation of chemotherapy to the date of the last follow-up or death.

REFERENCES:
- [Derived] Wu J, Zhang S, Yu S, An G, Wang Y, Yu Y, Liang L, Wang Y, Xu X, Xiong Y, Shao D, Shi Z, Li N, Wang J, Jin D, Liu T, Cui Y. Nivolumab plus anlotinib hydrochloride in advanced gastric adenocarcinoma and esophageal squamous cell carcinoma: the phase II OASIS trial. Nat Commun. 2024 Oct 15;15(1):8876. doi: 10.1038/s41467-024-53109-4. PMID 39406730